CLINICAL TRIAL: NCT02049385
Title: A Pathophysiological Study to Determine if Enhancing Glutamate Transporter Function Produces Antidepressant Effects in Patients With Major Depressive Disorder
Brief Title: Does Enhanced Glutamate Transporter Function Produce Antidepressant Effects in People With Major Depression?
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Severe side effects & lack of target engagement
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 140041; 14-M-0041 (Other: The National Institutes of Health)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-07

CONDITIONS: Depression
Keywords: Glutamate; Pathophysiology; Depression; Treatment
MeSH Terms: conditions — Depression | interventions — Diazoxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Diazoxide (Experimental): Subjects received 200-400 mg daily of diazoxide orally for three weeks; the dose was, adjusted depending on side effects and response.
  Interventions: Drug: Diazoxide
- Placebo (Experimental): Subjects received a matched placebo for three weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diazoxide — A nondiuretic vasodilator thiazide-related agent
  Arms: Diazoxide
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Background:

- At least one third of individuals with major depressive disorder (MDD) remain treatment-refractory after receiving currently available antidepressants underscoring the urgent need for new antidepressant therapies. Of the novel pharmacotherapeutic strategies seeking to rapidly alleviate depressive symptoms, glutamatergic modulators have emerged as promising potential targets. The present study sought to examine the potassium (KATP) channel activator diazoxide as a possible treatment for MDD. Diazoxide increases glutamate uptake from the synaptic cleft by activating the KATP channel to chronically increase expression of the excitatory amino acid transporter (EAAT)-2 system in glial cells. Diazoxide is FDA-approved for the treatment of sulfonylurea-induced hypoglycemia, hypoglycemia due to hyperinsulinemia, and hypertension.

Objectives:

- To assess the ability of diazoxide, potassium channel activator, to improve overall depressive symptomatology in patients with treatment-resistant MDD currently experiencing a major depressive episode. The efficacy of a three-week course of diazoxide will be compared to three weeks of placebo. The MADRS will serve as the main outcome measure

Eligibility:

- Adults 18 to 65 years old with MDD who are currently depressed without psychotic features.

Design:

* Study Phase I (Day -28 to 0):

  -- Screen and taper off medications (Days -28 to -14): Prior to consenting to this study, subjects will have undergone a screening consisting of laboratory tests, psychiatric and medical history, and psychiatric and physical examinations under protocol 01-M-0254, "The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Volunteers". After consenting to this study, patients will be tapered off medications. Medications allowed and not allowed are listed in Appendix 1. Patients will be reminded to report all drugs, OTC products, and other agents to the investigators so that they can screen to avoid interactions that might make participation unsafe or might confound the research results. Patients are expected to meet all inclusion and exclusion criteria before medications are tapered (which is usually 1-2 weeks long). Subjects who are not taking medications will enter the drug-free period directly. All participants must have a score of ≥20 on the MADRS at screening and baseline of Study Phase I. Subjects who do not have a score of ≥20 on the MADRS by the end of Study Phase I will be excluded and will receive standard treatment.
* Drug-free period (Day -14 to day 0):

  -- Subjects will begin a 2-week drug-free period prior to the administration of diazoxide or placebo.
* Study Phase II (Day 0 to 56):

  * In this study phase, subjects will be blindly randomized to receive either diazoxide 200-400 mg/day (given BID) or a placebo administered daily by mouth for three weeks. All patients except those who have a 50% or greater decrease in MADRS from baseline at the end of the first cross over point will cross over. To avoid carry-over effects between the different test sessions, there will be an interval of 14-21 days, pending response to test session 1. Subjects will then be blindly crossed over to the second experimental condition (either diazoxide or placebo) for another three weeks. All subjects who discontinue the study or who complete study phase II will then receive either clinical treatment or the opportunity to participate in another research protocol. Patients maintaining response to treatment condition 1 after two weeks will receive an additional one week washout before being crossed over to condition 2.The total duration of the study is approximately 11-13 weeks. The duration of Study Phase I including the 14-day drug-free period is approximately 4 weeks. Study phase II is 8-9 weeks long. Thus, the total duration of the study is approximately 11-13 weeks, except for those patients who were unmedicated at time of entry into the study and therefore do not need to undergo the initial tapering off medications. Subjects will be required to be hospitalized during the entire study. Passes will be permitted if the subject is clinically stable and the pass does not interfere with the study or unit procedures.

DETAILED DESCRIPTION:
Objective:

To date, available pharmacological treatments for major depressive disorder (MDD) have proven to be only modestly effective during the acute phase. We have been systematically testing different glutamatergic modulators in patients with mood disorders in order to develop improved therapeutics. A recent report found that the (beta)-lactam antibiotic ceftriaxone increased glutamate uptake by increasing GLT1(EAAT2) function and had antidepressant-like effects in animal models. Using the learned helplessness model of depression we developed outbred lines, defined a new anatomy of helplessness, and determined that synaptic loss due to excess extracellular glutamate appears to be involved in the pathophysiology of helplessness; these animals show a 40% decrease in EAAT2 astrocytic transporter expression. Together, these data suggest that astrocytic glutamate reuptake systems may be central to the pathophysiology and treatment of depression, and that agents that directly increase astrocytic glutamate uptake may represent a novel class of antidepressants.

With this protocol, we propose to test a specific new mechanism that uses diazoxide to chronically increase expression of the glutamate transporter EAAT2, resulting in removal of glutamate from the synaptic cleft. Diazoxide enhances glutamate uptake in glia by activating ATP-sensitive potassium (KATP) channels. We expect that this effect will reduce excessive glutamate transmission and be associated with acute antidepressant effects. The model presented here is a clinically testable one. If successful, it may lead to the development of a group of novel pharmacological treatments for major depressive disorder.

Study Population:

24 individuals with treatment-resistant major depressive disorder.

Design:

Male and female patients diagnosed with MDD, ages 18 to 65 years, currently experiencing a major depressive episode, will be recruited for this study. The study will comprise the double-blind crossover administration of either diazoxide (200-400 mg/day given orally) or placebo. The study will assess the efficacy of three weeks of a glutamate transporter enhancer (diazoxide, 200-400 mg/day given orally) compared with placebo in improving overall depressive symptomatology in patients with treatment-resistant MDD. Other aims of the study include: 1) determining whether changes in brain neurochemicals (glutamate) correlate with antidepressant response (as measured by decreases in Montgomery-Asberg Depression Rating Scale (MADRS) total scores) in response to diazoxide in patients with treatment-resistant MDD; and 2) examining other potential biomarkers of response.

Outcome Measures:

Primary: MADRS total score. Secondary outcome measures: proportion of subjects achieving remission (MADRS score less than or equal to 10) and response (more <50% reduction from baseline in MADRS total score); change from baseline in Beck Depression Inventory (BDI), Hamilton Anxiety Rating Scale (HAM-A), Hamilton Depression Rating Scale (HAM-D), Visual Analog Scale (VAS), and the Columbia Suicide Severity Rating Scale (C-SSRS) total scores.

ELIGIBILITY:
* INCLUSION CRITERIA:

  * 18 to 65 years of age.
  * Women of child bearing potential must have a negative serum pregnancy test and confirmed (by the investigator) use of two effective methods of contraception (see below).
  * Each subject must be capable of understanding all required tests and examinations and must sign an informed consent document.
  * Subjects must fulfill DSM-IV criteria for MDD, single episode or recurrent without psychotic features, based on clinical assessment and confirmed by a structured diagnostic interview (SCID-P). Subjects must be experiencing a current major depressive episode of at least four weeks duration.
  * Subjects must have an initial score of at least 20 on the MADRS at screening and at baseline of study Phase I.
  * Subjects must have a current or past history of lack of response to two adequate antidepressant trials (may be from the same chemical class) operationally defined using the modified-Antidepressant Treatment History Form (ATHF).

EXCLUSION CRITERIA:

* Current psychotic features or a current or past diagnosis of schizophrenia or any other psychotic disorder as defined in the DSM-IV.
* Subjects with a history of DSM-IV drug or alcohol dependency or abuse (except for caffeine or nicotine dependence) within the preceding three months.
* Head injury that results in loss of consciousness exceeding five minutes (for the imaging component of the study).
* Subjects with a DSM IV Axis II diagnosis of borderline or antisocial personality disorder.
* Pregnant or nursing women or women of child bearing potential not using two medically accepted means of contraception (including oral, injectable, or implant birth control, condoms, a diaphragm with spermicide; intrauterine devices (IUD); tubal ligation; abstinence; or partner with vasectomy).
* Serious, unstable medical illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
* Subjects with hyperthyroidism or clinical hypothyroidism.
* Subjects with one or more seizures without a clear and resolved etiology.
* Clinically significant abnormal laboratory tests (including blood glucose).
* Diabetes
* Fasting plasma glucose concentration >120 mg/dl
* Upright diastolic blood pressure <60mmHg on three occasions 30 minutes apart (based on scheduled research measurements).
* Treatment with a reversible MAOI within four weeks of study Phase II.
* Treatment with fluoxetine within five weeks of study Phase II.
* Treatment with any other disallowed concomitant medication 14 days before randomization.
* Treatment with clozapine or ECT within one month of randomization.
* Lifetime history of deep brain stimulation.
* Subjects who, in the investigator's judgment, pose a current serious suicidal or homicidal risk.
* Positive HIV test
* Contraindications to MRI (metal in body, claustrophobia, etc)

No structured psychotherapy will be permitted during the study.

Definition of treatment-resistance

All subjects are required to have previously failed to respond to two adequate antidepressant trials (may be from the same chemical class). Adequacy of antidepressant trials will be determined via the clinician administered modified ATHF.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01-03; Primary Completion 2016-07-21 (Actual); Study Completion 2016-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aitken RC. Measurement of feelings using visual analogue scales. Proc R Soc Med. 1969 Oct;62(10):989-93. doi: 10.1177/003591576906201005. No abstract available. PMID 4899510
- [Background] Akhondzadeh S, Mojtahedzadeh V, Mirsepassi GR, Moin M, Amini-Nooshabadi H, Kamalipour A. Diazoxide in the treatment of schizophrenia: novel application of potassium channel openers in the treatment of schizophrenia. J Clin Pharm Ther. 2002 Dec;27(6):453-9. doi: 10.1046/j.1365-2710.2002.00445.x. PMID 12472985
- [Background] Altamura CA, Mauri MC, Ferrara A, Moro AR, D'Andrea G, Zamberlan F. Plasma and platelet excitatory amino acids in psychiatric disorders. Am J Psychiatry. 1993 Nov;150(11):1731-3. doi: 10.1176/ajp.150.11.1731. PMID 8214185

RESULTS

PARTICIPANT FLOW:
Groups:
- Diazoxide, Then Placebo: Subjects received 200-400 mg daily of diazoxide orally for three weeks; the dose was adjusted depending on side effects and response.
- Placebo, Then Diazoxide: Subjects received a matched placebo for three weeks.
Period: First Intervention
Arm/Group | Diazoxide, Then Placebo | Placebo, Then Diazoxide
Started | 4 | 2
Completed | 1 | 2
Not Completed | 3 | 0
Period: Second Intervention
Arm/Group | Diazoxide, Then Placebo | Placebo, Then Diazoxide
Started | 1 | 2
Completed | 1 | 0
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Subjects received 200-400 mg daily of diazoxide orally for three weeks; the dose was, adjusted depending on side effects and response.
Arm/Group | All Participants
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: MADRS Change at Day 7
Description: Change in Montgomery Asberg Depression Rating Scale (MADRS) from baseline to 7 days post-treatment. The range of values is from 0 - 60, with a higher score indicating increased depressive symptoms. A score of 7-19 indicates mild depression; 20-34 indicates moderate depression; >34 indicates severe depression.
Time Frame: 7 days
Population: The analysis included those subjects who started treatment and completed treatment with Diazoxide or Placebo through at least 7 days.
Measure: Median (Full Range); unit: percentage of change in units of scale
Groups:
- Diazoxide: Subjects received 200-400 mg daily of diazoxide orally for three weeks; the dose was adjusted depending on side effects and response.
Arm/Group | Diazoxide | Placebo
Number analyzed (Participants) | 6 | 3
percentage of change in units of scale | 0 [0 to 100] | 10 [0 to 100]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Diazoxide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diazoxide (N=6) | Placebo (N=3)
Chest pain (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Discomfort (General disorders) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Weight increased (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Oedema (Metabolism and nutrition disorders) | 3 | 0
Chills (Musculoskeletal and connective tissue disorders) | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Akathisia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 0
Irregular sleep phase (Nervous system disorders) | 0 | 1
Poor quality sleep (Nervous system disorders) | 0 | 2
Sedation (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Decreased activity (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Irregular breathing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Dizziness (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
As only 1 participant completed both treatment arms, no formal statistical analysis of the primary outcome (MADRS) possible. Study halted due to severe side effects & lack of target (KATP channel) engagement measured by insulin sensitivity index.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes